CLINICAL TRIAL: NCT06102603
Title: Biobased Polyester Versus Synthetic Fiberglass Casts for Treating Stable Upper Limb Fractures in Children: a Randomized Controlled Trial
Brief Title: Biobased Polyester Versus Synthetic Fiberglass Casts for Treating Stable Upper Limb Fractures in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 110245-F
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-09

CONDITIONS: Upper Limb Fracture
Keywords: Pediatric upper limb fracture; casting; Bioabased polyester; Synthetic cast

STUDY DESIGN:
Intervention Model Description: The clinical trial was approved by the research ethics review committee of the author's hospital (Number XXX) and informed consent was obtained from the legal guardian of each patient. Between Feb 2022 and Nov 2022, all children (age range, 4-15 years) with radiography-diagnosed stable upper limb fractures (including radius, ulna, and distal humerus fractures such as Garland type I9 supracondylar fractures of the humerus) diagnosed at the orthopedic outpatient clinic or emergency room of a tertiary trauma center hospital were eligible for recruitment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the biobased polyester cast group (Experimental): biobased polyester cast was applied
  Interventions: Other: the biobased polyester cast
- the synthetic fiberglass cast group (Active Comparator): synthetic fiberglass cast was applied
  Interventions: Other: the synthetic fiberglass cast

INTERVENTIONS:
Other: the biobased polyester cast — long arm casting
  Arms: the biobased polyester cast group
Other: the synthetic fiberglass cast — long arm casting
  Arms: the synthetic fiberglass cast group

SUMMARY:
From Feb 2022 to Nov 2022, we undertook a single-center prospective randomized trial involving 100 children with cast-immobilized stable upper limb fractures. These patients were randomized into either biobased polyester or synthetic fiberglass groups. All patients were regularly followed up till the cast removal which occurred approximately 3-4 weeks after immobilizing. Objective clinical findings and subjective patient questionnaire were all collected and analyzed.

DETAILED DESCRIPTION:
The clinical trial was approved by the research ethics review committee of the author's hospital and informed consent was obtained from the legal guardian of each patient. Between Feb 2022 and Nov 2022, all children (age range, 4-15 years) with radiography-diagnosed stable upper limb fractures (including radius, ulna, and distal humerus fractures such as Garland type I supracondylar fractures of the humerus) [9] diagnosed at the orthopedic outpatient clinic or emergency room of a tertiary trauma center hospital were eligible for recruitment.

ELIGIBILITY:
Inclusion Criteria:

* stable upper limb fractures (including radius, ulna, and distal humerus fractures such as Garland type I supracondylar fractures of the humerus) diagnosed at the orthopedic outpatient clinic or emergency room of a tertiary trauma center hospital

Exclusion Criteria:

* displaced or unstable fractures indicated for close or open reduction and fixation
* previous surgeries to the affected upper limb
* history of any chronic skin pathology (e.g., atopic dermatitis)
* known allergy to cast materials

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
the number of patients with fracture union | one month after intervention
  clinical outcome
the number of complications | one month after intervention
  clinical outcome
patient satisfaction questionnaire | one month after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tsungyu Lan, Study Chair — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
the study protocol could be shared
Supporting Information: Study Protocol, SAP
Time Frame: one year

REFERENCES:
- [Derived] Lan TY, Chen CW, Huang YH, Lin SM, Liang CT, Chang CH, Rwei SP. Biobased polyester versus synthetic fiberglass casts for treating stable upper limb fractures in children: a randomized controlled trial. BMC Musculoskelet Disord. 2024 Jan 2;25(1):23. doi: 10.1186/s12891-023-07138-7. PMID 38166834